CLINICAL TRIAL: NCT05994144
Title: "Effectiveness of Video Observed Therapy in the Management of Tuberculosis"
Brief Title: "Conducting A Study On Video Observed Therapy In The Management Of Tuberculosis"
Acronym: VOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AISH7
Record Dates: First submitted 2023-07-19; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-05

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Digital health; video observed therapy; treatment adherence
MeSH Terms: conditions — Tuberculosis; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: For all participants who are randomised into VOT arm or traditional DOTS arm. Control group : Patients allocated into the traditional DOTS arm will follow the usual protocol as all other patients assigned to DOTS under Ministry of Health Malaysia Intervention group : Patient will be observed on their daily TB medication consumption via teleconference by using WhatsApp video call.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (No Intervention): The control group, traditional DOTS is the group who will be attending daily to their respective PR-1/PR-2 throughout intensive phase.
- INTERVENTION ARM (VOT) (Active Comparator): The intervention group, video observed therapy (VOT) is the group who will be teleconferencing daily with their respective PR-1/PR-2 TB team via WhatsApp throughout the intensive phase.
  Interventions: Other: VIDEO OBSERVED THERAPY

INTERVENTIONS:
Other: VIDEO OBSERVED THERAPY — Video-observed therapy is the usage of teleconferencing to observe anti-TB medication ingestion.
  Arms: INTERVENTION ARM (VOT)

SUMMARY:
The aim of this study is to measure the effectiveness usage of VOT in the treatment of TB in terms of treatment adherence. The study will be a randomized controlled trial and will involve 240 TB patients. The study is aimed to commence by December 2023. The study period will be for 4 months.

DETAILED DESCRIPTION:
There is an urgent need to produce an integrated e-health system in tackling the issue of remote monitoring for patient adherence. For example, in TB infection which requires close monitoring for better treatment outcomes. The usage of digital health products replacing the traditional DOTS will be a cost-effective method and will also bode convenient for patients and staff.

Video Observed Therapy (VOT) usage as the alternative digital health method replacing traditional DOTS will be more effective in tackling adherence issues. This method has already been tried in many countries like the United States of America (USA), the United Kingdom (UK), Italy, and Moldova, and has proven to be more effective than traditional DOTS.

For instance, a study by Story et al. reveals that a total of 70% of patients on VOT successfully completed ≥80% of a 2-month observation compared with only 31% of those on traditional DOTS (95% CI 3.10 to 9.68). A proposed intervention of adapting VOT in TB treatment is a practical move, as it can improve treatment compliance and also has the added benefit of being cost-effective.

1.4 Research Question What is the effectiveness of Video Observed Therapy (VOT) in the management of tuberculosis (TB) compared to the traditional Directly Observed Treatment Short Course Strategy (DOTS)?

1.5 Study Objectives

1.5.1 General Objective The general objective of this study is to compare the effectiveness of VOT with traditional DOTS in the management of TB.

1.5.2 Specific Objectives I. To develop VOT intervention in the management of TB. II. To compare the effectiveness of VOT as compared to traditional DOTS. III. To measure patient satisfaction using VOT.

ELIGIBILITY:
Inclusion Criteria:

i. All PTB smear-positive patients. ii. Patients aged 18 years and above. iii. Possess a digital phone or other equivalent gadget equipped with a WhatsApp application.

iv. Able to accurately identify each TB medication.

Exclusion Criteria:

i. Recurrent PTB infection. ii. Patients who are extremely ill, have no proper social support, no caretakers, and are hospitalized.

iii. Patients in prison during the time of diagnosis or treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment adherence in percentage from both arms | 60 days
  Number of days medicine consumed/over 60 days intensive period

SECONDARY OUTCOMES:
Seroconversion rate | 60 days
  Number of successful sero-conversion patients from sputum smear positive to sputum smear negative by the end of the intensive phase.
Side effects incidents report | 60 days
  Number of reported side effects detected from both arms.
Patients suffering with side effects | 60 days
  Number of patients having side effects detected from both arms.
Degree of patient's satisfaction | Questionnaire using Likert scale. "Score 1:least satisfied,Score 5: most satisfied"
  The degree of satisfaction of the participants from both arms.
Time save | 120 days
  Overall time spent by patients from both arms.
Cost saving | 60 days
  Overall money spent by patients from both arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sultanah Nur Zahira, Kuala Terengganu, Terengganu, Malaysia

IPD SHARING:
Plan to Share IPD: No
IPD WILL NOT BE SHARED FOR UNSPECIFIED REASONS